CLINICAL TRIAL: NCT04978025
Title: The Value of Colloidal Silver in the Treatment of COVID-19
Brief Title: Colloidal Silver, Treatment of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, PROFESSOR, Hôpital Universitaire Sahloul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: colloidal silver and COVID-19
Record Dates: First submitted 2020-11-05; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: SARS (Severe Acute Respiratory Syndrome)
Keywords: colloidal silver; treatment; COVID-19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — colloidal silver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver Group (Experimental): * Orally: the colloidal agent 1 dose of 30ml, 3 times a day for 5 days (use a plastic measuring cup and not a measuring cup or a metal spoon)
  * By inhalation: nebulization of 5ml of colloidal silver solution once, 3 times a day for 5 days.
  Interventions: Drug: Colloidal Silver
- Placebo Group (Placebo Comparator): * Orally: EPPI 1 dose of 30 ml, 3 times a day for 5 days
  * By inhalation: nebulization of 5ml of EPPI solution once a day, 3 times a day for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colloidal Silver — Orally: colloidal silver 1 dose of 30ml, 3 times a day for 5 days (use a plastic measuring cup and not a measuring cup or a metal spoon)
  and By inhalation: nebulization of 5ml of colloidal silver solution once, 3 times a day for 5 days.
  Other Names: Experimental
  Arms: Silver Group
Drug: Placebo — Orally: EPPI 1 dose of 30 ml, 3 times a day for 5 days By inhalation: nebulization of 5ml of EPPI solution once a day, 3 times a day for 5 days.
  Arms: Placebo Group

SUMMARY:
Noble metals such as gold and silver have been appreciated for millennia not only for their beauty but also for their ability to fight diseases.

Silver nanoparticles (AgNPs) have been employed as chemical drugs thanks to their unique physiochemical and chemical properties as well as biological features, such as anti-inflammatory, anti-angiogenesis, antiplatelet, antifungal, anti-cancer and antibacterial activities I

DETAILED DESCRIPTION:
Noble metals such as gold and silver have been appreciated for millennia not only for their beauty but also for their ability to fight diseases.

Silver nanoparticles (AgNPs) have been employed as chemical drugs thanks to their unique physiochemical and chemical properties as well as biological features, such as anti-inflammatory, anti-angiogenesis, antiplatelet, antifungal, anti-cancer and antibacterial activities Infectious diseases account for more than 20% of global mortality and viruses are responsible for about one-third of these deaths. Highly infectious viral diseases such as severe acute respiratory (SARS), Middle East respiratory syndrome (MERS) and coronavirus disease (COVID-19) are emerging more frequently and their worldwide spread poses a serious threat to human health and the global economy.

The current COVID-19 pandemic, caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) .

ELIGIBILITY:
Inclusion Criteria:

* Inclusion of any patient, over the age of 18, consulting the Sahloul emergencies, Sousse for symptoms of COVID -19 dating less than 10 days and having a positive COVID-19 on the PCR test and typical scanner.

Exclusion Criteria:

* Any pregnant or breastfeeding woman
* patient with an expectation of survival of less than 24 hours
* Dyspnea leading to heart failure
* Hepatic insufficiency
* Chronic respiratory failure
* Renal failure, clearance <20ml • min-1 • 1.73 • m-²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Chage of clinical status | 10 DAYS
  the distribution of clinical status assessed on the 7-point ordinal scale on day 10 of the study

SECONDARY OUTCOMES:
Adverse events | ON 1 month
  adverse events throughout the study period
the duration of hospitalization | ON 11 days
  number of days of hospitalization
the duration of the different respiratory assistance modes | ON 11 days
  the duration of the different respiratory assistance modes
all-cause mortality | ON 1 month
  the cause and the date of Death

CONTACTS AND LOCATIONS:
Overall Officials: Boukef Riadh, professor, Principal Investigator — HU Sahloul
Locations (1):
- HU Sahloul, sousse, Tunisia, Sousse, Itinéraire Ceinture Cité Sahloul, Tunisia

IPD SHARING:
Plan to Share IPD: No